CLINICAL TRIAL: NCT04498104
Title: Analysis of Personal Constructs in Borderline Personality Disorder and Its Relation With Severity and Therapeutic Outcome
Brief Title: Cognitive Conflict in Borderline Personality Disorder
Acronym: BPDCONFLICT
Status: Completed | Type: Observational
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Dr. Guillem Feixas, Professor, University of Barcelona
Other Study IDs: UBipcsBPD1
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Borderline Personality Disorder
Keywords: Repertory grid technique; Predictors of outcome; Implicative dilemma; Dilemmatic construct; Personal Construct Theory
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Borderline Personality Disorder: Borderline personality disorder diagnosed participants
  Interventions: Other: Psychological assessment
- Control: Healthy participants
  Interventions: Other: Psychological assessment

INTERVENTIONS:
Other: Psychological assessment — Psychological assessment with the repertory grid technique (RGT) in order to quantify cognitive conflicts.

SUMMARY:
Background: Borderline personality disorder (BPD) is a severe psychological condition characterized by emotional, interpersonal and self-image instability in addition to impulsive behaviour. Although there have been several explanatory models and psychotherapy approaches that have been designed to comprehend and intervene on BPD, most seem not to recognize idiosyncratic cognitive conflict as an important feature on this disorder. Adding personal dilemmas, such as those conceptualized in personal construct theory, as a key element to BPD's explanatory model could provide a better picture to understand this disorder and possibly to enhance effectiveness of current psychotherapy approaches. Despite the fact that constructivist explanatory models have been used and tested in several clinical populations, there is little work done studying the relevance of inner conflicts in BPD. According to the prototypical symptomatology manifested by these patients, psychological instability can be assumed as a transversal feature present in this disorder; therefore, a larger amount of cognitive conflict can be expected in BPD patients.

Method and Analysis: In order to test this assumption, this study aims to examine the characteristics of the interpersonal cognitive system of patients diagnosed with BPD and note their potential differences with the general population using the repertory grid technique, a complex assessment tool derived from personal construct theory. Statistical analyses will be performed to examine whether the clinical sample tends to present with more cases and with higher number of cognitive conflicts than the control group. Likewise, the association between cognitive conflict and symptom severity will be explored. Results will be a first step to determine if cognitive conflicts have an important role in the explanation of BPD. This will also help to value the convenience to further investigate the efficacy of conflict resolution psychotherapy interventions with these patients. This research work is undertaken in the context of a funded predoctoral research program.

DETAILED DESCRIPTION:
Out of all personality disorders, BPD is one of the most life-threatening and psychological distressful due the symptomatic manifestation of impulsive behavior along with emotional, interpersonal and self-image instability. Suicidality and Non-Suicidal Self-Injury (NSSI) rates in this population are extremely high, and worrying for the families and mental health professionals. Over the last decades, BPD has obtained broad attention and many psychological treatments have been proposed to deal with its main symptoms. Although some treatments have been proven to be empirically effective in some domains, clearly not all experienced symptoms are successfully targeted, and some cases seem not to be helped even when treated by the more efficacious approaches. Perhaps, the explanatory models from which these psychotherapies emerge could have underestimated important aspects such as personal dilemmas.

Cognitive conflict has been defined and conceptualized by different psychological orientations, but only a few have included this phenomenon as an influential factor in the understanding of the origin and nature of psychological disorders and their psychotherapy proposals. Those that have considered inner conflicts have mainly focused on theoretical based dilemmas the academics would perceive relevant or common instead of exploring potential ideographic conflicts patients may have.

Being a disorder that is noticeably characterized by identity disturbances, finding relevant unresolved cognitive conflicts regarding self and others in these patients is expected. Addressing these issues could be potentially useful to further develop an explanatory model for this disorder as well as to increase therapeutic resources to help with these unattended potential necessities.

The central aim of this research is to assess cognitive conflicts in BPD diagnosed individuals to determine their role in the explanatory model of this disorder. These findings would permit the consideration of adapting a dilemma-focused intervention module which could complement existing treatments for these patients. In addition, exploring other characteristics of self-construction and the construction of others that are assessed with the RGT would be of interest. The specific objectives of this study are:

1. To test the hypothesis that patients with BPD present more cognitive conflicts (i.e., implicative dilemmas and dilemmatic constructs) than a general population sample.
2. To explore the content of cognitive conflicts in patients with BPD.
3. To examine whether presence and/or frequency of cognitive conflicts is associated with severity of emotional symptoms in BPD patients.
4. To explore whether the presence and number of cognitive conflicts has any capacity to predict treatment outcome.
5. To examine the relevance of other aspects of the construction of the self and others to explain the psychological functioning of patients with a BPD diagnosis.

The hypothesis of this study are:

1. The percentage of participants with implicative dilemmas and/or dilemmatic constructs will be superior in the group of patients diagnosed with BPD compared to a control group (community sample).
2. The number of implicative dilemmas and/or dilemmatic constructs will be higher in the BPD group than in the control group.
3. Presence and higher number of cognitive conflicts will be associated with greater levels of general clinical symptomatology (such as depression, anxiety, etc.).
4. Presence and higher number of individual cognitive conflicts will predict poor treatment outcome one year after the initial assessment.

For exploratory purposes, the content of implicative dilemmas and dilemmatic constructs will be studied, as well as the differences with the control group regarding self-construction measures (self-ideal discrepancy, self-others discrepancy, ideal-others discrepancy) and other characteristics of the construction system (interpersonal cognitive differentiation and polarization) and its association with other clinical and sociodemographic variables.

ELIGIBILITY:
INCLUSION CRITERIA

* Aged between 18 and 60 years old.
* Having been diagnosed with BPD by a well-trained professional according to DSM-5 criteria.

EXCLUSION CRITERIA

* Having been diagnosed with bipolar disorder, psychotic disorder, prevalent continued and active substance abuse, disabling physical illness, organic cerebral dysfunctions or mental developmental severe difficulties.
* Not able to communicate either in Spanish or Catalan.
* Presence of other comorbid conditions such as other personality disorders, anxiety disorders, eating disorders, depression or non-disabling physical illness, will not be an exclusion motive, but will be recorded for statistical control purposes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study Population: The borderline personality group will be formed by participants diagnosed with BPD that receive treatment from outpatient or inpatient public and private mental health facilities in the local area of Barcelona, Spain (CSMA Benito Menni, ITA - especialistas en salud mental and ITLímit).
  The control group will be formed by healthy volunteers of a student sample from the University of Barcelona and a nonstudent community sample who were not receiving psychotherapy when evaluated. These participants will be matched by age, gender and educational level with the clinical sample.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Implicative dilemma | Through study completion, an average of 2 years.
  The repertory grid technique (RGT) is a personalized assessment procedure using a structured interview designed to make explicit the personal constructs (bipolar dimensions of subjective meaning) used to interpret and organize reality. An implicative dilemma can be identified when an individual does not perform a desired change due to the negative implications involved for their desired identity. The RGT can detect personal constructs in which the current perception of the self is similar to the ideal self (congruent constructs) and the constructs in which the subject's self-perception is contrary to their ideal construction (discrepant construct). A statistical analysis of the RGT reveals when a potential pole shift of a discrepant construct involves the pole shift of a congruent construct due to an existing association between the two constructs. Implicative dilemmas may cause dissatisfaction and psychological discomfort.
Dilemmatic construct | Through study completion, an average of 2 years.
  Dilemmatic constructs can be identified when an individual is not sure how would they like to be in a certain identity aspect. This type of cognitive conflict can be assessed and analyzed with the RGT in order to identify self-construction domains in which the person may find it difficult to choose how to ideally be. Indecision in regard to identity can add psychological distress to those who experience it.

SECONDARY OUTCOMES:
Diagnostic Interview for Borderlines - Revised (DIB-R) | Through study completion, an average of 2 years.
  It is a structured interview that helps to identify the potential presence of BPD by assessing 22 common statements for BPD patients. It explores aspects related to affectivity, cognition, impulsivity patterns and interpersonal relationships. The test provides an overall score from 0 to 10 that determines presence or absence of BPD (6 or higher indicates presence).
Structured Clinical Interview for DSM-IV-II (SCID-II) | Through study completion, an average of 2 years.
  It is a structured assessment interview aimed to identify the potential presence or absence of the personality disorders defined by the DSM-IV criteria. After completion, results show how many diagnostic criteria are met by the interviewee for each of the 13 personality disorder assesed. When evaluating BPD, scores can go from 0 to 9 (5 or higher indicates presence).
Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM) | Through study completion, an average of 2 years.
  It is a self-report questionnaire formed by 34 items (18 in the reduced version) that aims to assess the clinical state of the person in the following four dimensions: subjective well-being, problem/symptoms, general functioning and risk. All scales and an overall measure are computed in order to obtain scores that rank from 0 to 4 (higher scores indicates worse outcome).
Depression Anxiety Stress Scales (DASS-21) | Through study completion, an average of 2 years.
  It is a questionnaire created to quickly evaluate levels of depression, anxiety and stress. Respondents must score in a scale from 0 to 3 to describe the intensity or frequency they experienced about 21 different clinical symptoms during the previous week. Punctuations oscillate between 0 and 63 (higher scores indicates worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Feixas, Professor, Principal Investigator — University of Barcelona
Locations (3):
- Spain (3):
  - ITA - especialistas en salud mental, Barcelona
  - CSMA Bennito Menni - (Germanes Hospitalaries), Barcelona
  - ITLimit, Sant Cugat del Vallès

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Feixas G, Saul LA, Avila-Espada A. Viewing Cognitive Conflicts as Dilemmas: Implications for Mental Health. J Constr Psychol. 2009 Apr;22(2):141-169. doi: 10.1080/10720530802675755. Epub 2009 Feb 18. PMID 22629109
- [Background] Montesano A, Lopez-Gonzalez MA, Saul LA, Feixas G. A review of cognitive conflicts research: a meta-analytic study of prevalence and relation to symptoms. Neuropsychiatr Dis Treat. 2015 Dec 4;11:2997-3006. doi: 10.2147/NDT.S91861. eCollection 2015. PMID 26675503
- [Background] Feixas G, Compan V. Dilemma-focused intervention for unipolar depression: a treatment manual. BMC Psychiatry. 2016 Jul 12;16:235. doi: 10.1186/s12888-016-0947-x. PMID 27406383
- [Background] Feixas G, Bados A, Garcia-Grau E, Paz C, Montesano A, Compan V, Salla M, Aguilera M, Trujillo A, Canete J, Medeiros-Ferreira L, Soriano J, Ibarra M, Medina JC, Ortiz E, Lana F. A DILEMMA-FOCUSED INTERVENTION FOR DEPRESSION: A MULTICENTER, RANDOMIZED CONTROLLED TRIAL WITH A 3-MONTH FOLLOW-UP. Depress Anxiety. 2016 Sep;33(9):862-9. doi: 10.1002/da.22510. Epub 2016 Apr 22. PMID 27103215
- [Background] Feixas G, Paz C, Garcia-Grau E, Montesano A, Medina JC, Bados A, Trujillo A, Ortiz E, Compan V, Salla M, Aguilera M, Guasch V, Codina J, Winter DA. One-year follow-up of a randomized trial with a dilemma-focused intervention for depression: Exploring an alternative to problem-oriented strategies. PLoS One. 2018 Dec 13;13(12):e0208245. doi: 10.1371/journal.pone.0208245. eCollection 2018. PMID 30543642
- [Background] Paz C, Montesano A, Winter D, Feixas G. Cognitive conflict resolution during psychotherapy: Its impact on depressive symptoms and psychological distress. Psychother Res. 2019 Jan;29(1):45-57. doi: 10.1080/10503307.2017.1405172. Epub 2017 Nov 26. PMID 29173128
- [Background] Feixas G, Saul LA. The Multi-Center Dilemma Project: an investigation on the role of cognitive conflicts in health. Span J Psychol. 2004 May;7(1):69-78. doi: 10.1017/s1138741600004765. PMID 15139250
- [Background] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- See also: Link to our research group webpage "Intervention in Clinical and Health Psychology" — http://www.ub.edu/ipcs/es/